CLINICAL TRIAL: NCT06976229
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, and Preliminary Efficacy of Human Allogeneic Induced Pluripotent Stem Cell (iPSC)-Derived Motor Neuron Progenitor Cells (XS228 Cell Injection) in Patients With Subacute Spinal Cord Injury
Brief Title: Safety and Early Efficacy of iPSC-Derived Motor Neuron Progenitor Cells (XS228) in Subacute Spinal Cord Injury: A Phase I Trial
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: XellSmart Bio-Pharmaceutical (Suzhou) Co., Ltd. (Industry)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XS228-Allo-SCI-CN1-P01
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury; Safety; Clinical Trials; Efficacy; Induced Pluripotent Stem Cells; Human Motor Neuron Progenitor; Transplantation
Keywords: spinal cord injury; safety; efficacy; clinical trials; Induced Pluripotent Stem Cells; Human motor neuron progenitor; Transplantation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XS228 for injection (Experimental): The Single Ascending Dose (SAD) and Muliple Ascending Dose (MAD) stages were built up in the study. XS228 in SAD and MAD following intrathecal injection through lumbar puncture in Subacute Spinal Cord Injury participants.
  Interventions: Biological: Allogeneic Human Induced Pluripotent Stem Cell (iPSC)-Derived Motor Neuron Progenitor Cells

INTERVENTIONS:
Biological: Allogeneic Human Induced Pluripotent Stem Cell (iPSC)-Derived Motor Neuron Progenitor Cells — Description:
  The Single Ascending Dose (SAD) and Muliple Ascending Dose (MAD) stages were built up in the study. XS228 in SAD and MAD following intrathecal injection through lumbar puncture in subacute spinal cord Injury participants.For SAD,the participants will single intrathecal injection with the dose level as 5×10^7 cells 、1.5×10^8 cells. For MAD, the participants will intrathecal injection of XS228 in Day 1, Day15, Day 29, Day 43 under the dose level of 5×10^7 cells、1.5×10^8 cells.Dose escalation followed a rule-based 3+3 design.
  XS228 is an investigational, allogeneic cell therapy product composed of motor neuron progenitor cells (MNPCs) derived from human induced pluripotent stem cells (iPSCs). This advanced therapy medicinal product (ATMP) is being developed for the treatment of subacute spinal cord injury and represents a novel approach in regenerative medicine.
  Other Names: XS228 Cell Injection; XS228

SUMMARY:
This Phase I clinical trial is designed to evaluate the safety, tolerability of XS228 ( iPSC-Derived Motor Neuron Progenitor Cells) in patients with Subacute Spinal Cord Injury

ELIGIBILITY:
Inclusion Criteria:

Age: 18 to 65 years (inclusive), regardless of gender.

Etiology: Cervical (C4) to lumbar (L2) spinal cord injury (SCI) caused by traumatic injury or surgery-related factors.

Severity:

Classified as ASIA Impairment Scale (AIS) Grades A, B, or C. MRI-confirmed evidence of spinal cord injury.

Disease Stage:

Primary SCI occurring 14 to 60 days prior to screening (subacute phase).

Contraception:

Participants of childbearing potential (male and female) must agree to use effective non-hormonal contraceptive methods during the trial and for 6 months after trial completion.

Compliance:

Voluntarily participate in the clinical study. Ability to understand and comply with study procedures. Participant or legal guardian can provide written informed consent.

Exclusion Criteria:

* Neurological Inability

Primary spinal cord injury (SCI) during screening with concomitant severe traumatic brain injury precluding neurological function assessment.

Respiratory/Circulatory Instability

High cervical SCI (C1-C3) causing respiratory/circulatory compromise requiring endotracheal intubation or tracheostomy.

Life-Threatening Multiorgan Dysfunction

Concurrent severe injuries to other organ systems with life-threatening dysfunction.

Unstable Thoracoabdominal Injuries

Injuries to lungs, liver, kidneys, spleen, etc., deemed unstable by the investigator.

Prior Spinal Pathology

History of SCI or coexisting spinal disorders (e.g., ankylosing spondylitis, spinal deformities, primary/metastatic spinal tumors, spinal vascular malformations, syringomyelia).

Local Infection/Increased ICP

Active infection at the lumbar puncture site or intracranial hypertension during screening.

Severe Infections

Sepsis, septic shock, or severe pneumonia (per IDSA/ATS 2007 diagnostic criteria).

Confounding Neurological/Psychiatric Conditions

Parkinson's disease, severe dementia, myasthenia gravis, stroke, Guillain-Barré syndrome, diabetic neuropathy, or other conditions interfering with study assessments.

Cardiac Abnormalities (any of the following):

Congestive heart failure (NYHA Class III/IV). Severe uncontrolled arrhythmias (e.g., sick sinus syndrome, third-degree AV block).

Unstable angina or acute myocardial infarction within 3 months prior. Pulmonary Complications

Pulmonary hypertension, pulmonary embolism, or suspected embolism during screening.

Uncontrolled Hypertension/Hypotension

Systolic BP >160 mmHg or diastolic BP >100 mmHg; or systolic BP <90 mmHg or diastolic BP <60 mmHg.

Active Autoimmune Diseases

Requiring immunosuppressants (e.g., uncontrolled hyperthyroidism, systemic lupus erythematosus).

Immunosuppressant Non-Compliance

Unwillingness or inability to use immunosuppressants per protocol.

Laboratory Abnormalities (any of the following):

ALT/AST >2×ULN or total bilirubin >2×ULN. eGFR <60 mL/min/1.73m² (CKD-EPI 2021 formula). APTT/PT >2.5×ULN (without anticoagulants). Platelets <100×10⁹/L or hemoglobin <90 g/L. Allergy

History of severe allergies or hypersensitivity to trial drug/excipients (human albumin, lactated Ringer's solution).

Infectious Diseases

HBsAg+ with HBV DNA >1000 IU/mL; HCV-Ab+; HIV-Ab+; or TP-Ab+. Lumbar Puncture Refusal

Unwillingness to undergo intrathecal administration procedures. Pregnancy/Lactation

Females who are pregnant or breastfeeding. Malignancy

Active malignancy or anticancer therapy within 5 years prior. Recent Clinical Trial Participation

Enrollment in another drug trial within 3 months prior. Investigator Discretion

Any condition deemed unsuitable for participation by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2028-02-21 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events (AEs) and serious adverse events (SAEs) | 28 days after administration in the SAD treatment and 28 days after the final (fourth) administration in the MAD treatment
  To evaluate the safety and tolerability of XS228 in A single dose and the last dose of MAD treatment of Subacute Spinal Cord Injury through Adverse events (AE) related to XS228 ,incidence of SAE（serious adverse events).The severity of AEs observed during the trial will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
DLT（Dose-limiting toxicity） | 28 days after administration in the SAD treatment and 28 days after the final (fourth) administration in the MAD treatment
  To evaluate the safety and tolerability of XS228 in A single dose and the last dose of MAD treatment of Subacute Spinal Cord Injury through DLT（Dose-limiting toxicity）.A DLT is defined as any Grade 3 or higher adverse event (based on NCI-CTCAE Version 5.0) that occurs within 28 days following single-dose administration in the SAD treatment or the final dose in the MAD treatment ， which is assessed as related to XS228, or any other significant adverse event as determined by the Safety Review Committee (SRC) .
RP2D（Recommended Phase 2 Dose） | After the last participant in the MAD treatment of the Phase I trial completes the 28-day DLT observation period
  After the last participant in the MAD treatment of the Phase I trial completes the 28-day DLT observation period following their final dose, the Safety Review Committee (SRC) and the sponsor will jointly determine the recommended dose for Phase II based on safety and preliminary efficacy data from Phase I.

SECONDARY OUTCOMES:
Improvement in ASIA Impairment Scale (AIS) grade | Improvement in ASIA Impairment Scale (AIS) grade from baseline at Day 29, Day 90, Day 180, Day 270, and Day 360 after the first dose administration.
  To evaluate the Improvement in ASIA Impairment Scale (AIS) grade after the administration 0f XS228(ASIA Impairment Scale (AIS) grade)
Changes in American Spinal Injury Association (ASIA) Motor Score | From baseline at Day 29, Day 90, Day 180, Day 270, and Day 360 after the first dose administration.
  Changes in motor scores assessed by the ASIA score scale (total score range from 0 to 100, higher values represent a better outcome)
Changes in American Spinal Injury Association (ASIA) Sensory Score | From baseline at Day 29, Day 90, Day 180, Day 270, and Day 360 after the first dose administration.
  Changes in sensory scores assessed by the ASIA score scale (total score range from 0 to 224, higher values represent a better outcome)
Changes in Spinal Cord Independence Measure-III (SCIM-III) | From baseline at Day 29, Day 90, Day 180, Day 270, and Day 360 after the first dose administration.
  SCIM-III(range: 0-100, with lower score indicating greater disability)

CONTACTS AND LOCATIONS:
Overall Officials: Limin Rong, prof and M.D, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, the sponsor has not yet finalized a decision regarding the sharing of individual participant data (IPD). The potential risks and benefits of data sharing, including patient privacy, regulatory requirements, and intellectual property considerations, are still under evaluation. A final determination will be made following further internal review and alignment with applicable data protection laws, institutional policies, and ethical guidelines. If IPD sharing is approved in the future, details regarding data accessibility, anonymization methods, and request procedures will be specified in an updated plan.